CLINICAL TRIAL: NCT00147277
Title: ADVANCE-D: ATP Delivery for Painless ICD Therapy
Brief Title: ADVANCE-D: Antitachycardia Pacing (ATP) Delivery for Painless Implantable Cardioverter Defibrillator (ICD) Therapy
Acronym: ADVANCE_D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 900AD
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Results first posted 2009-05-12 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2015-08

CONDITIONS: Tachycardia, Ventricular; Ventricular Fibrillation
Keywords: ATP; Thachy; FVT
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8 pulses (Active Comparator): 8 pulses Anti-Tachycardia Pacing (ATP) delivered in the right ventricle to treat Fast Ventricular Tachycardia (FVT)
  Interventions: Device: Implantable Cardiac Defibrillator
- 15 pulses (Experimental): 15 pulses Anti-Tachycardia Pacing (ATP) delivered in the right ventricle to treat Fast Ventricular Tachycardia (FVT)
  Interventions: Device: Implantable Cardiac Defibrillator

INTERVENTIONS:
Device: Implantable Cardiac Defibrillator — Medtronic Marquis Family ICD, capable of Anti Tachy Pacing (ATP) for Fast Ventricular Tachycardia (FVT) via Ventricular Fibrillation (VF) zone

SUMMARY:
The purpose of this study is to estimate and quantify the difference in efficacy of two sequences of ATP therapies (burst 15 pulses, 88% versus burst 8 pulses, 88%) during an episode of spontaneous rhythms classified as fast ventricular tachycardia (FVT) via ventricular fibrillation (VF) in patients who have a Class I or II A indication for ICD implantation, and thus to promote the "painless" therapy aspect of ICD treatment and improve quality of life outcomes for patients.

DETAILED DESCRIPTION:
Main objective: Compare & quantify efficacy of two different sequences of burst ATP strategies for the termination of ventricular tachycardia (with Cycle Lenght (CL) of 240ms-320ms) from baseline to 12 months post randomisation in patients who are treated with ATP -8 pulses, 88% versus patients who are treated with ATP -15 pulses, 88%

Secondary objectives:

* Estimate the efficacy of ATP in successfully treating FVT episodes for patients in primary and secondary prevention
* Estimate acceleration rate or degeneration of ATP therapy for treating spontaneous FVT episodes in the ATP 15 vs 8 arm
* Compare the likelihood of syncopal events associated with spontaneous FVT episodes
* Estimate the percent reduction in number of shocks delivered per patient for treating spontaneous FVT episodes
* Evaluate different possible predictors of ATP success: VT rate, underlying disease, Anti-Arrhythmic Drugs (AAD), infarct zone, etc.

ELIGIBILITY:
Inclusion Criteria:

* ICD indications (Class I-II A) according to the guidelines (patient with coronary artery disease [CAD] or non-CAD in primary or secondary ICD prevention)
* Patients have been implanted with a Medtronic Marquis family ICD capable of ATP for FVT via VF

Exclusion Criteria:

* Patient's life expectancy less than 1 year due to a non-cardiac chronic disease
* Patient on heart transplant list which is expected in < 1 year
* Patient's age less than 18 years
* ICD replacements and upgrading (single chamber [SC] ICD® dual chamber [DC] ICD)
* Unwillingness or inability to provide written informed consent
* Enrollment in, or intention to participate in, another clinical study during the course of this study
* Inaccessibility for follow-up at the study center
* Ventricular tachyarrhythmias associated with reversible causes
* Brugada syndrome, long QT and hypertrophic cardiomyopathy (HCM) patients
* Other electrical implantable devices (neurostimulators, etc.)
* Mechanical tricuspid valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 925 (Actual)
Dates: Start 2004-03; Primary Completion 2006-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Lunati, Dr., Principal Investigator — Ospedale Niguarda Cà Granda - Milano; Riccardo Cappato, Dr., Principal Investigator — Istituto Policlinico S. Donato Milanese; Massimo Santini, Prof., Principal Investigator — San Filippo Neri - Roma; Angel Arenal, Dr., Principal Investigator — Hospital Gregorio Marañón, Madrid; Josè Luis Merino, Dr., Principal Investigator — Hospital Universitario La Paz; Arcadio Garcia-Alberola, Dr., Principal Investigator — Hospital Universitario Virgen de la Arrixaca; Johann Mermi, Dr., Principal Investigator — Clinic Center Dortmund; Pascal Defaye, Dr., Principal Investigator — University Hospital, Grenoble
Locations (1):
- Medtronic Italia SpA, Sesto San Giovanni, MI, Italy

REFERENCES:
- [Background] Lunati M, Defaye P, Mermi J, Garcia-Alberola A, Merino JL, Arenal A, Cappato R, Navarro X, Passardi M, Santini M. Improvement of quality of life by means of antitachy pacing: from PainFREE to the ADVANCE-D Trial. Pacing Clin Electrophysiol. 2006 Dec;29 Suppl 2:S35-9. doi: 10.1111/j.1540-8159.2006.00488.x. PMID 17169131

RESULTS

PARTICIPANT FLOW:
Groups:
- 8 Pulses Anti-Tachycardia Pacing (ATP): 8 pulses ATP delivered in the right ventricle to treat Fast Ventricular Tachycardia (FVT)
- 15 Pulses Anti-Tachycardia Pacing (ATP): 15 pulses ATP delivered in the right ventricle to treat Fast Ventricular Tachycardia (FVT)
Period: Overall Study
Arm/Group | 8 Pulses Anti-Tachycardia Pacing (ATP) | 15 Pulses Anti-Tachycardia Pacing (ATP)
Started | 475 | 450
Completed | 475 | 450
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 8 Pulses Anti-Tachycardia Pacing (ATP) | 15 Pulses Anti-Tachycardia Pacing (ATP) | Total
Number analyzed (Participants) | 475 | 450 | 925
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 214 | 203 | 417
  >=65 years | 261 | 247 | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.9) | 63.4 (12.2) | 63.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 48 | 114
  Male | 409 | 402 | 811
Region of Enrollment [Number; unit: participants]
  Italy | 180 | 169 | 349
  Germany | 109 | 106 | 215
  France | 84 | 77 | 161
  Spain | 76 | 75 | 151
  Portugal | 7 | 8 | 15
  Belgium | 8 | 7 | 15
  Israel | 9 | 6 | 15
  United Kingdom | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Anti Tachycardia Pacing (ATP) Therapy to Terminate Fast Ventricular Tachycardia (With Cycle Length of 240ms-320msec)
Description: Termination of Ventricular Tachycardia is calculated as percentage of successfully terminated episodes, adjusted for multiple events with (GEE) method. This technique yields an average therapy efficacy and 95% CI that is based on number of patients, number of episodes per patient, and magnitude of the correlation between responses within patients.
Time Frame: one year
Population: 934 patients were created in the electronic data capture system, only 925 patients were enrolled in the study: 4 patients in the 8 pulses arm and 5 patients in the 15 pulses arm were created by mistake and excluded from analysis. The analysis were performed with the Intention To Treat (ITT) method.
Measure: Number; unit: Percentage of FVT episodes terminated
Arm/Group | 8 Pulses Anti-Tachycardia Pacing (ATP) | 15 Pulses Anti-Tachycardia Pacing (ATP)
Number analyzed (Participants) | 475 | 450
Percentage of FVT episodes terminated | 64.9 | 69.7

2. Secondary Outcome: Efficacy of ATP in Successfully Treating FVT for Patients in Primary and Secondary Prevention
Time Frame: one year
Reporting Status: Not Posted

3. Secondary Outcome: Acceleration Rate or Degenerated Into VF of ATP for Treating FVT in the 2 Arms
Time Frame: one year
Reporting Status: Not Posted

4. Secondary Outcome: Percent Reduction in Shocks Delivered Per Patient for Treating FVT
Time Frame: one year
Reporting Status: Not Posted

5. Secondary Outcome: Compare Likelihood of Syncopal Events Associated With FVT
Time Frame: one year
Reporting Status: Not Posted

6. Secondary Outcome: Evaluate Different Possible Predictors of ATP Success
Time Frame: one year
Reporting Status: Not Posted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No